CLINICAL TRIAL: NCT02276287
Title: HIV Positive Patient's Cognitive and Emotional Illness Perception: a Possible Tool for Understanding Adherence?
Brief Title: HIV Patients Illness Perception and Adherence
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Daniela Leone, PsyD, MS, research fellow, University of Milan
Other Study IDs: UMilan
Record Dates: First submitted 2014-10-23; First posted 2014-10-28 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: HIV
Keywords: Adherence; HAART; HIV; Illness Perception; IPQ-R

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: the study aimed to explore HIV positive patients' perceptions toward illness and treatment, and their associations with demographic and clinical variables, in particular with adherence.

Methods: the study was conducted at the outpatients clinic of Infectious Disease of a University Hospital in the north of Italy. Patients were asked to fill out the Illness Perception Questionnaire-Revised. Patient's adherence was measured by: viral load (HIV-RNA copies/ml) and presence at the check up.

DETAILED DESCRIPTION:
Data collection Participants were recruited in the waiting room, before their check up visit or the blood test; a researcher explained them the aim of the study and asked them a written informed consent to participate. The accepting patients were asked to fill out the Illness Perception Questionnaire Revised (IPQ-R). Demographic, clinical and adherence data were also collected.

Measures:

1. Demographic and clinical data: demographic information included age, gender, marital status, education, employment status, nationality. Clinical information, extracted from participants' medical records, included: years diagnosed with HIV, patient history of antiretroviral therapy (ART), years of therapy, presence of fix dose combination of antiretroviral drugs, current therapeutic regimen's type, total number of pills per day, presence of other drugs' therapies, HIV acquisition risk.
2. Illness representations: measured with the Italian validate version of the IPQ-R24. The questionnaire is divided in three sections: 1) disease identity; 2) opinions and 3) causes. While items on disease identity have dichotomous responses (yes/no), items regarding opinions and causes are constituted by a 5 points Likert scale (from "1=completely disagree" to "5=completely agree").

   Identity section explores patients' beliefs about the disease's nature. Fourteen symptoms are listed and patients have to indicate if they have experienced them since being diagnosed with the disease and, if so, if they believe that their symptoms are linked to the disease or not. Opinions section is composed by 38 items exploring how, at the moment, patients perceive their illness condition. Items are grouped into seven factors: 1) Timeline (perception of chronic vs acute duration); 2) Cyclical symptoms (perception of a cyclic vs stable disease); 3) Consequences (perception that the disease has or not serious physical, psychological and social consequences on patients' life); 4) Personal control (perceptions that actions can or cannot be taken to effectively manage the disease); 5) Treatment control (high or low trust in the treatment and its efficacy); 6) Coherence (high or low understanding of the disease); 7) Emotional responses (prevalence of negative emotions vs positive).

   Causes section lists 18 possible illness causes and patients have to rate their level of agreement with each item as a cause of their disease.
3. Adherence indexes : measured by HIV-RNA copies/ml and presence at the check up visits(scheduled every 3 months). Patients were considered "adherent" in case of: undetectable viral load or HIV-RNA <40 copies/ml and regular presence at the check up visits (≤ 3 months). Adherence indexes were collected only for patients under treatment (naïve patients and patients in therapy from <1 month were excluded).

Data analysis Descriptive statistics were used for demographic and clinical characteristics, IPQ-R data and adherence outcomes. Data were analyzed using SPSS® version 21.0 for Windows.

Independent t-tests, one-way ANOVA with LSD post hoc multiple comparisons tests and Pearson correlational analysis were used for the analysis of demographic/clinical variables and IPQ-R Identity and Opinion continuous variables. Mann-Whitney U-test and Kruskal-Wallis Chi-Squared test were used on IPQ-R Cause ordinal variables.

One-way ANOVA with LSD post hoc multiple comparisons tests were also used to compare means between the adherence indexes and IPQ-R Identity and Opinion continuous variables. Kruskal-Wallis Chi-Squared tests were used on IPQ-R Cause ordinal variables. Values of p ≤0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. HIV positivity
2. age ≥18 years
3. to be able to understand and provide informed consent
4. to be able to understand a questionnaire in Italian
5. not to be psychiatric patient
6. not to be alcohol and/or drugs' abuser

Exclusion Criteria:

1. not HIV positive patients
2. age <18 years
3. inability to understand and provide informed consent
4. inability to understand a questionnaire in Italian
5. to be psychiatric patient
6. to be alcohol and/or drugs' abuser

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV positive patients recruited at the outpatients clinic of Infectious Disease, S.Paolo University Hospital, Milan, Italy during their check up visit or blood test
Sampling Method: Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Illness representations | participants will be followed for the duration of their hospital access, an expected average of 2 hours
  Illness Perception Questionnaire Revised (IPQ-R)

SECONDARY OUTCOMES:
demographic data | participants will be followed for the duration of their hospital access, an expected average of 2 hours
  age, gender, marital status, education, employment status, nationality
clinical data | from date of HIV diagnosis until the date of the visit in which patients were recruited for the study , assessed from 1984 to 2014
  years diagnosed with HIV, patient history of antiretroviral therapy, years of therapy (first therapy and current therapy), presence of fix dose combination of antiretroviral drugs, current therapeutic regimen's type (once a day and twice a day), total number of pills per day, presence of other drugs' therapies, HIV acquisition risk.
Adherence | Adherence indexes assessed at the last check up visit (from 2 weeks up to 12 months)
  HIV-RNA copies/ml, and presence at the check up visits

CONTACTS AND LOCATIONS:
Overall Officials: Elena Vegni, Professor, Study Director — University of Milan